CLINICAL TRIAL: NCT01256177
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL) Extended Release as Monotherapy in the Treatment of Patients With Bipolar Depression
Brief Title: Evaluate the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL) Extended Release as Monotherapy in the Treatment of Patients With Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D144CC00005
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; Mental disease,
MeSH Terms: conditions — Bipolar Disorder; Mental Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Quetiapine Fumarate (SEROQUEL) Extended Release
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine Fumarate (SEROQUEL) Extended Release — Quetiapine fumarate extended release(XR) will be administered orally, once daily in the evening. The initial dose will be 50 mg. This dose will be adjusted on Day 2 to 100 mg, on Day 3 to 200 mg, and on Day 4 to 300 mg and after.
  Arms: 1
Drug: Placebo — Placebo matching quetiapine extended release(XR) 50 mg, 200 mg, and 300 mg tablets will be orally administered once daily, in the evening. The initial dose will be 50 mg. This dose will be adjusted on Day 2 to 100 mg, on Day 3 to 200 mg, and on Day 4 to 300 mg and after.
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the superior efficacy of quetiapine extended release(XR) mono-therapy, administered once daily compared to placebo, in the treatment of depressive symptoms in patients with Bipolar I and Bipolar II Disorder

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male and female patients, aged 18 to 65 years, inclusive.
* Meets Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) criteria for bipolar disorder I or bipolar II, most recent episode depressed (296.5x and 296.89x).
* Hamilton Rating Scale for Depression (HAM-D) (17-item) total score of ≥ 20 and HAM-D item 1 (depressed mood) score ≥ 2 at enrolment and randomisation.
* Patients must be able to understand and comply with the requirements of the study,as judged by the Investigator

Exclusion Criteria:

* Patients with a current Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) diagnosis other than bipolar disorder
* Patients whose Young Mania Rating Scale (YMRS) total score >12 at enrolment and randomisation.
* Patients with >8 mood episodes during the past 12 months at enrolment.
* Patients whose current episode of depression exceeds 12 months or is less than 4 weeks from enrolment.
* Patients with a history of non-response to an adequate treatment (6 weeks) with more than 2 classes of antidepressants during their current episode.
* Alcohol or other substance dependence or abuse as defined by Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) criteria at enrolment that is not in extended full or extended partial remission (12 months or longer), except caffeine and nicotine dependence.
* Patients who, in the Investigator's judgment, pose a current serious suicidal or homicidal risk, have a Hamilton Rating Scale for Depression (HAM-D) item 3 score ≥ 3, or have made a suicide attempt within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuxin Gu Niufan, MD, Principal Investigator — Shanghai Mental Health Center- Peking University sixth Hospital; Dhaval Desai, Study Director — Wilmington, DE - Delaware; Frank Hou, Study Chair — Astrazeneca China
Locations (12):
- China (12):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an

REFERENCES:
- [Derived] Li H, Gu N, Zhang H, Wang G, Tan Q, Yang F, Ning Y, Zhang H, Lu Z, Xu X, Shi J, Gao C, Li L, Zhang K, Tian H, Wang X, Li K, Li H, Xu Y, Xie S, Yu X. Efficacy and safety of quetiapine extended release monotherapy in bipolar depression: a multi-center, randomized, double-blind, placebo-controlled trial. Psychopharmacology (Berl). 2016 Apr;233(7):1289-97. doi: 10.1007/s00213-016-4215-z. Epub 2016 Feb 25. PMID 26911380
- See also: D144CC00005_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1804&filename=D144CC00005_Clinical_Trial_Disclosure_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 56-days (8 week), multicenter, double-blind, randomized, parallel group, Phase III study was done to compare the efficacy and safety of quetiapine XR with placebo in the treatment of patients with bipolar depression. In total 296 patients were randomized in 19 centers in the China between December 2010 and November 2012.
Pre-assignment Details: 361 patients were enrolled in the study of which 296 patients were randomized and 65 patients were not randomized. Reasons for patients not being randomized are (22 due to eligiblity criteria not fullfilled, 40 due to subject decision, 3 due to others).
Groups:
- Placebo: Placebo matching Quetiapine XR.
- Quetiapine XR: Quetiapine Fumarate (SEROQUEL) Extended Release Tablet administered orally, once daily in the evening.
Period: Overall Study
Arm/Group | Placebo | Quetiapine XR
Started | 148 | 148
Completed | 98 | 111
Not Completed | 50 | 37
Not completed — Withdrawal by Subject | 23 | 22
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 8 | 9
Not completed — Severe Non-Compliance to Protocol | 4 | 2
Not completed — Condition under Investigation Worsened | 1 | 0
Not completed — Lack of Efficacy | 11 | 2
Not completed — TG=593mg/dL, not fit to participate. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) Of the 148 patients randomized to each group, 1 in each group did not receive treatament. In addition, there were 15 patients (7 placebo; 8 quetiapine XR) for which no MADRS data were collected. All 17 patients are included in the Reason Not Completed Section above.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine XR | Total
Number analyzed (Participants) | 140 | 139 | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.8 (11.0) | 33.4 (11.9) | 33.1 (11.4)
Age, Customized [Number; unit: Participants]
  18 - 39 years | 105 | 102 | 207
  40 - 65 years | 35 | 37 | 72
Sex/Gender, Customized [Number; unit: Participants]
  Female | 73 | 72 | 145
  Male | 67 | 67 | 134
Race/Ethnicity, Customized [Number; unit: Participants] — Race, Asian Ethnicity, Chinese
  Participants
    Race,Asian | 140 | 139 | 279
    Ethnicity, Chinese | 140 | 139 | 279
Weight [Mean (Standard Deviation); unit: Kilogram (Kg)] | 65.2 (12.3) | 63.8 (13.5) | 64.5 (12.9)
MADRS total score at baseline [Mean (Standard Deviation); unit: Scores on a scale] — Montgomery-Asberg Depression Rating Scale (MADRS) total score range: 0 to 60, the higher the score, the more severe.
  Scores on a scale | 28.8 (5.3) | 28.5 (5.4) | 28.6 (5.3)
Bipolar Diagnosis [Number; unit: Participants] — Bipolar - I disorder is characterized by one or more manic or mixed episodes, usually alternating with major depressive episodes.
  Bipolar - II disorder is characterized by one or more major depressive episodes and at least one hypomanic episode.
  Participants
    Bipolar - I | 72 | 70 | 142
    Bipolar - II | 68 | 69 | 137
Rapid cycling course [Number; unit: Participants] — Rapid cycling course defined as ≥ 4 mood episodes in the past year.
  Participants
    No | 132 | 134 | 266
    Yes | 8 | 5 | 13
Duration of present depressive episode [Mean (Standard Deviation); unit: Weeks] | 12.3 (10.0) | 13.7 (10.3) | 13 (10.1)
Years since Bipolar diagnosis [Mean (Standard Deviation); unit: Years] | 3.2 (4.7) | 2.8 (4.6) | 3 (4.6)
Attempted sucide [Number; unit: Participants]
  No | 124 | 128 | 252
  Yes | 16 | 11 | 27
Hamilton Rating Scale for Depression (HAM-D) total score at baseline [Mean (Standard Deviation); unit: Scores on a scale] — HAM-D total score range: 0 to 53, the higher the score, the more severe.
  Scores on a scale | 23.2 (3.0) | 23.5 (3.6) | 23.3 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 2) to End of Study (Week 8) in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS total score range: 0 to 60, the higher the score, the more severe, Change : Total MADRS score at week 8 minus score at baseline
Time Frame: Baseline to Week 8
Population: Full Analysis Set (Number of participants at Week 8: Placebo=100; Quetiapine XR=114)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Scores on a scale
  Change from Baseline to End of Study | -15.27 (0.81) | -18.48 (0.78)
  Baseline | 28.8 (0.45) | 28.5 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 8 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures (MMRM); Baseline MADRS total value as covariate, treatment, bipolar strata, visit, treatment-visit interaction as fixed effects and centre as random; Least Square Mean difference vs Placebo = -3.22, 95% CI 2-sided [-5.39 to -1.04], Standard Error of Mean 1.10

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score Response (Subjects With ≥50% Reduction From Baseline to Week 8 in MADRS Total Score)
Description: Montgomery-Asberg Depression Rating Scale (MADRS) total score range: 0 to 60, the higher the score, the more severe, Response was defined as ≥50% reduction in MADRS total score from baseline
Time Frame: 8 weeks from baseline
Population: Full Analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Participants | 62 | 93
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds ratio was modeled by logistic regression adjusted for centre, baseline score, and bipolar strata; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.56 to 4.13] — Quetiapine XR/Placebo

3. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score Remission (the Proportion of Subjects With a MADRS Total Score ≤ 12 at Week 8 Assessment)
Description: Montgomery-Asberg Depression Rating Scale (MADRS) total score range: 0 to 60, the higher the score, the more severe, Remission was defined as MADRS total score ≤12
Time Frame: After 8 week of start of treatment
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Participants | 59 | 88
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds ratio was modeled by logistic regression adjusted for centre, baseline score, and bipolar strata; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.46 to 3.86] — Quetiapine XR/Placebo

4. Secondary Outcome: Change From Baseline to Each Assessment in MADRS Total Score
Description: MADRS total score range: 0 to 60, the higher the score, the more severe.
Time Frame: Baseline to Week 8
Population: Full Analysis Set (Number of participants at each assessment : Baseline (Placebo=140, Quetiapine XR= 139), Week 1 (Placebo=140, Quetiapine XR= 139), Week 2 (Placebo=127, Quetiapine XR= 128), Week 4 (Placebo=114, Quetiapine XR= 120), Week 6 (Placebo=102, Quetiapine XR= 114), Week 8 (Placebo=100, Quetiapine XR= 114)).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Scores on a scale
  Change from Baseline to Week 1 | -4.14 (0.50) | -5.62 (0.51)
  Change from Baseline to Week 2 | -7.70 (0.64) | -10.13 (0.65)
  Change from Baseline to Week 4 | -11.05 (0.69) | -14.18 (0.69)
  Change from Baseline to Week 6 | -13.96 (0.76) | -16.04 (0.74)
  Change from Baseline to Week 8 | -15.27 (0.81) | -18.48 (0.78)
  Baseline | 28.8 (0.45) | 28.5 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 1 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.029, Mixed Model Repeated Measure (MMRM); [statistical method as in outcome 1, analysis 1]; Least Square Mean difference vs Placebo = -1.47, 95% CI 2-sided [-2.79 to -0.15], Standard Error of Mean 0.67
Statistical Analysis 2: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 2 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measure (MMRM); [statistical method as in outcome 1, analysis 1]; Least Square Mean difference vs Placebo = -2.43, 95% CI 2-sided [-4.16 to -0.69], Standard Error of Mean 0.88
Statistical Analysis 3: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 4 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.001, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 1, analysis 1]; Least Square Mean difference vs Placebo = -3.12, 95% CI 2-sided [-5.00 to -1.25], Standard Error of Mean 0.95
Statistical Analysis 4: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 6 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.045, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 1, analysis 1]; Least Square Mean difference vs Placebo = -2.08, 95% CI 2-sided [-4.12 to -0.05], Standard Error of Mean 1.03
Statistical Analysis 5: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 8 in MADRS total score based on observed cases (OC); Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 1, analysis 1]; Least Square Mean difference vs Placebo = -3.22, 95% CI 2-sided [-5.39 to -1.04], Standard Error of Mean 1.10

5. Secondary Outcome: Change From Baseline to Week 8 in HAM-D Total Scores
Description: HAM-D total score range: 0 to 53, the higher the score, the more severe. Change : Total HAM-D score at week 8 minus score at baseline
Time Frame: Baseline to Week 8
Population: Full Analysis Set (Number of Participants at Week 8: Placebo=100; Quetiapine XR=114).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Scores on a scale
  Change from Baseline to Week 8 | -12.92 (0.61) | -15.16 (0.59)
  Baseline | 23.2 (1.96) | 23.5 (1.87)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 8 in HAM-D total score based on observed cases (OC); Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures (MMRM); Baseline HAM-D total value as covariate, treatment, bipolar strata, visit, treatment-visit interaction as fixed effects and centre as random; Least Square Mean difference vs Placebo = -2.24, 95% CI 2-sided [-3.88 to -0.61], Standard Error of Mean 0.83

6. Secondary Outcome: Change From Baseline to Week 8 Assessment in the Clinical Global Impression Bipolar - Severity (CGI-BP-S)
Description: CGI-BP severity of illness-Overall bipolar range = 1-7, the higher is the total score,the more severe is the disease. CGI-BP severity of illness-Depression range: 1-7, the higher is the total score, the more severe is the disease
Time Frame: Baseline to Week 8
Population: Full Anlaysis Set (Number of Participants at Week 8: Placebo=100; Quetiapine XR=112)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Scores on a scale
  CGI-BP-S score for Overall Bipolar (BP) Illness | -1.73 (0.12) | -2.24 (0.12)
  CGI-BP-S score of depression | -1.81 (0.13) | -2.28 (0.13)
  CGI-BP-S overall score Baseline | 4.5 (.065) | 4.6 (.067)
  CGI-BP-S score for depression Baseline | 4.5 (.065) | 4.6 (.068)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Change from baseline to Week 8 assessment in the CGI-BP-S score for overall Bipolar (BP) illness based on observed cases (OC); Test type: Superiority or Other; p = 0.003, Mixed Model Repeated Measures (MMRM); Baseline CGI-BP-S score for overall BP illness as covariate, trt, bipolar strata, visit, trt-visit interaction as fixed effect and centre as random; Least Square Mean difference vs Placebo = -0.51, 95% CI 2-sided [-0.84 to -0.17], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 8 assessment in the CGI-BP-S score of depression based on observed cases (OC); Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures (MMRM); Baseline CGI-BP-S score for depression as covariate, trt, Bipolar strata, visit, trt-visit interaction as fixed effects and centre as random; Least Square Mean difference vs Placebo = -0.47, 95% CI 2-sided [-0.81 to -0.13], Standard Error of Mean 0.17

7. Secondary Outcome: The Proportion of Patients at Week 8 With a Clinical Global Impression - Bipolar - Change (CGI-BP-C) of "Much" or "Very Much" Improved
Description: Clinical Global Impression - Bipolar - Change (CGI-BP-C) of "much" or "Very much" improved is defined as a change in CGI-BP overall bipolar illness score ≤ 2 where 1 = very much improved, 2 = much improved.
Time Frame: After 8 weeks of start of treatment
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Participants | 65 | 91
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds ratio between treatment groups was modeled by logistic regression adjusted for centre, baseline score and bipolar Strata; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.26 to 3.36] — Quetiapine XR/Placebo

8. Secondary Outcome: Change From Baseline to Week 8 in Item 10 of Montgomery-Asberg Depression Rating Scale (MADRS) for Suicidal Ideation
Description: MADRS item 10 (suicidal ideation) score range: 0 to 6, the higher the score, the more severe, Change: MADRS item 10 score at week 8 minus score at baseline
Time Frame: Baseline to Week 8
Population: Full Analysis Set (Number of Participants at Week 8: Placebo=100; Quetiapine XR=114)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Scores on a scale
  Change from Baseline to Week 8 | -0.76 (0.06) | -0.98 (0.06)
  Baseline | 1.2 (.094) | 1.0 (.083)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Change from Baseline to Week 8 in MADRS item 10 score for suicidal ideation based on observed cases (OC); Test type: Superiority or Other; p = 0.005, Mixed Model Repeated Measures (MMRM); Baseline MADRS item 10 score as covariate, treatment, bipolar strata, visit, treatment-visit interaction as fixed effect and centre as random; Least Square Mean difference vs Placebo = -0.22, 95% CI 2-sided [-0.38 to -0.07], Standard Error of Mean 0.08

9. Secondary Outcome: Incidence of Treatment-emergent Mania (AE of Mania or Hypomania, Defined as Young Mania Rating Scale [YMRS] Score ≥16 on 2 Consecutive Assessments or Final Assessment)
Description: The incidence of treatment-emergent mania is defined as ≥16 of YMRS total score on 2 consecutive assessments or at final assessment, YMRS total score range: 0-60, the higher is the total score the more severe is the disease.
Time Frame: After 8 weeks of start of treatment
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Quetiapine XR
Number analyzed (Participants) | 140 | 139
Participants | 4 | 1
Statistical Analysis 1: Comparison: Placebo vs Quetiapine XR; Test type: Superiority or Other; p = 0.233, Regression, Logistic; Odds ratio between treatment groups was modeled by logistic regression adjusted for centre, strata and baseline score; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.03 to 2.38] — Quetiapine XR/Placebo

ADVERSE EVENTS:
Description: Full Analysis Set (FAS) Of the 148 patients randomized to each group, 1 in each group did not receive treatment.
Arm/Group | PLACEBO | QUETIAPINE XR
Serious Adverse Events (participants affected / at risk) | 3/147 | 0/147
Other Adverse Events (participants affected / at risk) | 43/147 | 81/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=147) | QUETIAPINE XR (N=147)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=147) | QUETIAPINE XR (N=147)
CONSTIPATION (Gastrointestinal disorders) | 4 (5) | 17 (17)
DRY MOUTH (Gastrointestinal disorders) | 7 (7) | 21 (22)
NAUSEA (Gastrointestinal disorders) | 10 (10) | 3 (3)
FATIGUE (General disorders) | 2 (3) | 13 (14)
NASOPHARYNGITIS (Infections and infestations) | 10 (10) | 3 (3)
DIZZINESS (Nervous system disorders) | 16 (19) | 29 (30)
SOMNOLENCE (Nervous system disorders) | 11 (11) | 36 (36)
INSOMNIA (Psychiatric disorders) | 12 (14) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish or present any such results until the earlier of (i) the date of the first Study results publication, or in case of a Multi-Centre Study the first Multi-Centre Results publication, authorized by AstraZeneca and (ii) the end of the eighteen (18) month period following the completion, or early termination, of the Study at all participating sites.